CLINICAL TRIAL: NCT06688916
Title: A Comprehensive Assessment of Altered Embodiment in Individuals With Spinal Cord Injury
Acronym: SCI_Embodiment
Status: Recruiting | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2024-13
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injuries (SCI)
Keywords: spinal cord injury; embodiment; bodily sensations; magnetic resonance imaging; daily life
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Individuals with SCI - Behavioral assessment: 15 individuals with SCI will perform a comprehensive behavioral assessment of embodiment (see "Interventions"). A clinical assessment of sensory-motor symptoms will also be carried out.
  Interventions: Behavioral: Behavioral assessment
- Individuals with SCI - Behavioral assessment and fMRI: 25 individuals with SCI will perform a comprehensive behavioral assessment of embodiment and neural correlates of embodiment will be explored by means of an fMRI procedure (see "Interventions"). A clinical assessment of sensory-motor symptoms will also be carried out.
  Interventions: Behavioral: Behavioral assessment; Behavioral: Functional Magnetic Resonance Imaging (fMRI)
- Healthy controls - Behavioral assessment: 15 healthy controls will perform a comprehensive behavioral assessment of embodiment (see "Interventions").
  Interventions: Behavioral: Behavioral assessment
- Healthy controls - Behavioral assessment and fMRI: 25 individuals with SCI will perform a comprehensive behavioral assessment of embodiment and neural correlates of embodiment will be explored by means of an fMRI procedure (see "Interventions").
  Interventions: Behavioral: Behavioral assessment; Behavioral: Functional Magnetic Resonance Imaging (fMRI)

INTERVENTIONS:
Behavioral: Behavioral assessment — A comprehensive behavioral assessment of embodiment and its effect on daily living, taking into account pain, interoception, emotions and anxiety, sleep quality, life satsfaction and cognition.
Behavioral: Functional Magnetic Resonance Imaging (fMRI) — Neural mechanisms of embodiments will be explored with MRI sequences including structural MRI, resting-state and task-based fMRI of the head.
  The task will be a modified version of the rubber hand illusion, previously used to asess embodiment. Participants will be required to lay in the MRI with their legs bended upright and a screen placed at the level of their hips, which will show a pair of legs. The participant's leg will be stroked with a paintbrush while the image on the screen will be showing the virtual legs being stroked. Participants will be required to report how strongly they perceive the virtual legs as their own, as a measure of embodiment.
  Groups: Healthy controls - Behavioral assessment and fMRI; Individuals with SCI - Behavioral assessment and fMRI

SUMMARY:
Spinal cord injury (SCI) occurs when trauma or other factors damage the spinal cord, disrupting the flow of sensory information from the body to the brain. This interruption can interfere with embodiment-the body awareness and physical sensations processed by the brain-sometimes leading to a phenomenon called disembodiment.

For people with SCI, disembodiment may appear as unusual body sensations, like feeling that a limb is in a different position than it actually is. Such changes in body awareness can impact daily life, mental health, and rehabilitation outcomes.

Despite its importance, the study of embodiment in SCI remains limited. This project aims to explore how SCI alters embodiment, focusing on its specific characteristics, the effects on daily life, and the underlying brain activity as measured by functional magnetic resonance imaging (fMRI). Both people with and without SCI will participate.

Procedure: Participants will complete a single examination lasting 2 to 2.5 hours, including approximately 55 minutes in the MRI scanner (with preparation and follow-up).

ELIGIBILITY:
Inclusion Criteria for all participants:

* Age between 18 and 60
* Normal or corrected-to-normal visual acuity
* German or Italian native speaker

Additional Inclusion Criteria only for individuals with SCI:

* Diagnosis of traumatic spinal cord injury
* Lesion level below T1 (first thoracic vertebra)
* Time since injury >= 12 months
* Residual sensation on the upper leg (sensory capability of 1 or higher on at least one leg in the dermatomes L2 and L3 for both light touch and pin prick).

Exclusion Criteria for all participants:

* Pregnancy or breastfeeding
* Diagnosis of other psychiatric or neurological disorders (e.g. epilepsy, tumor in the central nervous system)
* Confirmed diagnosis of alcohol and/or drug abuse with active consumption within the last 6 months
* Confirmed diagnosis of traumatic brain injury, intended as visible changes in the brain diagnosed by a radiologist
* Stroke
* Inability to perform study procedures (e.g. inability to consent)

Additional Exclusion Criteria for both HC and SCI undergoing the fMRI procedure:

* Active medical devices (e.g. cardiac pacemaker)
* Inability to perform study procedures (e.g. claustrophobia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with spinal cord injury and healthy controls.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Score on the Body Feelings and Illusions questionnaire (BoFI) | Baseline
  A questionnaires that assess different dimensions of embodiment and disembodiment.

SECONDARY OUTCOMES:
Brain activity | Baseline
  Brain activity defined as changes in oxygen levels in the blood during the execution of the embodiment task, and at rest.
Strenght of the embodiment illusion | Baseline
  Strenght of the embodiment illusion during the fMRI procedures, measured through a Likert scale.
Qualitative assessment of embodiment | Baseline
  Qualitative assessment of the experience of embodiment by means of a semi-structured interview.
Score on the WHO Disability Assessment Scale (WHODAS-II) | Baseline
  A scale that assesses activity limitation and participation restriction in the daily life due to disability.
Pain severity | Baseline
  Intensity of pain measured on a visual analogue scale.
Score on the Positive and Negative Affect Schedule (PANAS) | Baseline
  A scale which measures positive and negative sensations over the course of the last week.
Anxiety score on the Hospital Anxiety and Depression Scale (HADS) | Baseline
  A scale the assesses the presence and the intensity of anxiety and depressive symptoms.
Depression score on the Hospital Anxiety and Depression Scale (HADS) | Baseline
  A scale the assesses the presence and the intensity of anxiety and depressive symptoms.
Score on the Pittsburgh Sleep Quality Index | Baseline
  A questionnaire assessing the quality of sleep.
Score on the Multidimensional Assessment of Interoceptive Awareness (MAIA) | Baseline
  A questionnaire assessing interoceptive awarness.
Score on the Inclusion of Others in the Self test (IOS) | Baseline
  A questionnaire assessing the relationship of the individual self with other entities (e.g., the body, the famiy, the society).
Score on the Montreal Cognitive Assessment (MoCA) | Baseline
  A test assessing cognitive functions such as memory, attention, language, and executive functions.
Score on the Satisfaction with Life Scale (SLS) | Baseline
  A scale assessing satisfaction in life.
Motor symptoms severity | Baseline
  Motor symptoms severity (from level A to E) based on the International Standards for Neurological Classification of spinal cord injury (ISNCSCI)
Demographics | Baseline
  Demographic information such as age, sex and education level, as well as time since injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Research, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No
The investigators plan to save anonymized data into public repositories. However, due to the size of the imaging data, a final decision has not yet been made.